CLINICAL TRIAL: NCT01838486
Title: Bladder Thermal Distention for Patients With Interstitial Cystitis / Painful Bladder Syndrome
Acronym: IC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 37/12
Record Dates: First submitted 2013-04-19; First posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Interstitial Cystitis; Painful Bladder Syndrome
Keywords: Interstitial cystitis; painful bladder syndrome; bladder hydrodistention; hyperthermia
MeSH Terms: conditions — Cystitis, Interstitial; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bladder Thermal Distention (BTD) (Experimental): Continuous irrigation of the bladder with warm saline (up to 45 Celsius) using the PelvixTT system
  Interventions: Procedure: Bladder Thermal Distention

INTERVENTIONS:
Procedure: Bladder Thermal Distention — Bladder Thermal Distention (BTD) is an approved procedure in Europe and Israel. Continuous irrigation of the bladder with warm saline with the PelvixTT system. The procedure will be performed on an outpatients basis. The procedure lasts 1 hour.
  Other Names: PelvixTT - Hyperthermia Elmedical LTD, Israel

SUMMARY:
Patients with Interstitial Cystitis / PBS will be treated with bladder thermal distention (BTD).

DETAILED DESCRIPTION:
In this study we will evaluate the efficacy of bladder thermal distention (BTD) in patients with IC/PBS.

Patients with previous failed conventional treatment (intravesical DMSO) will be recruited.

ELIGIBILITY:
Inclusion Criteria:

-All patients with interstitial cystitis / painful bladder syndrome (IC/PBS) who had previous intravesical treatment with DMSO

Exclusion Criteria:

* Active infection
* Urethral stricture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
o'leary sant questionnaire | up to 1 year
  o'leary sant questionnaire is a validated specific tool for evaluation of IC/PBS symptoms

SECONDARY OUTCOMES:
Bladder diary | up to 1 year
  symptoms like urgency. frequency and functional voided volumes will be monitored

CONTACTS AND LOCATIONS:
Overall Officials: Kobi Stav, MD, Principal Investigator — Assaf Harofe Medical Center
Locations (1):
- Assaf Harofe Medical Center, Ẕerifin, Israel